CLINICAL TRIAL: NCT01387451
Title: Cross Sectional Study on the Detection and Factors of Brown Adipose Tissue in Different Locations of Adults
Brief Title: The Detection and Factors of Brown Adipose Tissue in Different Locations of Adults
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Yiming Li, huashan Hospital
Other Study IDs: KY2010-115
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2010-04

CONDITIONS: Obesity
Keywords: Brown adipose tissue; Different regions; Chinese adults
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Adipose tissue, plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Retrospective studies have combined positron-emission tomography and computed tomography (PET-CT) to identify adipose tissue with a high rate of uptake of 18F-fluorodeoxyglucose(18F-FDG) as active brown adipose tissue(BAT). In addition, biopsy specimens and immunohistochemical staining with a UCP1-specific antiserum were used to indicate that normal adults were able to have BAT. However,these studies only chose few subjects and limited to the neck tissue. Therefore, the investigators intend to test BAT in different parts of adults and analyse the clinical factors.

DETAILED DESCRIPTION:
The investigators will promote the cross-sectional study from 2010 to 2013 in Shanghai. Data on demographic statistics, medical history,physical examination and fasting blood sample will be collected for all patients. Adipose tissue of adults will be collected from different regions, such as cervical, perirenal, along the large blood vessels and trachea, because they are included in the range of surgical therapy and are the major locations of BAT. Adipose tissue samples will be used to immunohistochemical stain, to detect the expression of BAT related genes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent surgical therapy and the operation scope includes BAT sample sites.

Exclusion Criteria:

* Pregnant women
* With implantable medical electronic instrument
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent surgical therapy from 2010 to 2013 in Huashan Hospital and the operation scope includes brown adipose tissue sample sites.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Doctor, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China